CLINICAL TRIAL: NCT04184440
Title: The Hypoglycemic Effect of Cyclocarya Paliurus Extract on Hyperglycemic Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QQLY2019
Record Dates: First submitted 2019-11-21; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Hyperglycemia
Keywords: Cyclocarya paliurus extract; hyperglycemia; pre-diabetes and diabetes
MeSH Terms: conditions — Hyperglycemia; Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Participants will be divided randomly into three groups，among which the intervention will start and end simultaneously.
Who Masked: Participant, Outcomes Assessor
Masking Description: The allocation of three groups is completed by the primary researcher,and unknown to participants and other reachers. It is the same in the size,color,shape and taste of capsules administrated by three groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator): corn starch；capsule，2 g/day，2 times/day；3 months
  Interventions: Dietary Supplement: placebo
- Cyclocarya paliurus extract (Experimental): aqueous extract of Cyclocarya paliurus；capsule，2 g/day，2 times/day；3 months
  Interventions: Dietary Supplement: Cyclocarya paliurus extract
- Cyclocarya paliurus compounds (Experimental): mixed aqueous extract of Cyclocarya paliurus and other traditional Chinese herbal medicines including Astragalus propinquus Schischkin，Dioscorea oppositifolia L.，Dendrobium nobile Lindl.，Salvia miltiorrhiza Bge. and Inulin；capsule，2 g/day，2 times/day；3 months
  Interventions: Dietary Supplement: Cyclocarya paliurus compounds

INTERVENTIONS:
Dietary Supplement: Cyclocarya paliurus extract — The participants are divided randomly into three groups，one of which are asked to Cyclocarya paliurus extract for three months .
  Arms: Cyclocarya paliurus extract
Dietary Supplement: Cyclocarya paliurus compounds — The participants are divided randomly into three groups，one of which are asked to take Cyclocarya paliurus compounds for three months .
  Arms: Cyclocarya paliurus compounds
Dietary Supplement: placebo — The participants are divided randomly into three groups，one of which are asked to take placebo for three months .
  Arms: placebo

SUMMARY:
This is a randomized double-blind controlled trial，aiming to investigate the hypoglycemic effect of Cyclocarya paliurus extract and Cyclocarya paliurus compounds on hyperglycemic populations without modifying their original treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* pre-diabetic or type 2 diabetic patients who are treated with only one oral antidiabetic agent and whose fasting plasma glucose is lower than 8.4 mmol;
* age:20-65 years;
* BMI :20-35kg/m2.

Exclusion Criteria:

* type 1 diabetic patients;
* type 2 diabetic patients with insulin treatment；
* pregnant or lactating women；
* adverse effect on intervention；
* acute or chronic inflammatory conditions;
* severe hepatic,kidney or other complications;
* other situations ineligible to intervention.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
changes of FPG | at 0 week，4th week and 12th week in the intervention period
  fasting plasma glucose
changes of HbA1c | at 0 week，4th week and 12th week in the intervention period
  glycated hemoglobin
changes of fasting insulin | at 0 week，4th week and 12th week in the intervention period
changes of OGTT | at 0 week，4th week and 12th week in the intervention period
  oral glucose tolerance test

SECONDARY OUTCOMES:
changes of blood lipids | at 0 week，4th week and 12th week in the intervention period
  total cholesterol，high density lipoprotein cholesterol，low density lipoprotein cholesterol，triglyceride
changes of gut microbiota | at 0 week，4th week and 12th week in the intervention period
  16s RNA sequencing
changes of short chain fatty acids | at 0 week，4th week and 12th week in the intervention period
  metabolites of microbiota in feces

CONTACTS AND LOCATIONS:
Locations (1):
- Shiyan Taihe Hospital, Shiyan, Hubei, China

IPD SHARING:
Plan to Share IPD: No